CLINICAL TRIAL: NCT00387049
Title: Anxiety Sensitivity Program for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Ruth Farrell/Associate Vice President, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA018734 (NIH); R01DA018734 (NIH)
Record Dates: First submitted 2006-10-10; First posted 2006-10-12 (Estimated); Last update posted 2010-10-22 (Estimated); Status verified 2006-10

CONDITIONS: Smoking Cessation
Keywords: Anxiety Sensitivity
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anxiety-specific smoking cessation care (Experimental)
  Interventions: Behavioral: Anxiety Sensitivity Program for Smoking Cessation
- Standard smoking cessation care (Active Comparator)
  Interventions: Behavioral: Anxiety Sensitivity Program for Smoking Cessation

INTERVENTIONS:
Behavioral: Anxiety Sensitivity Program for Smoking Cessation

SUMMARY:
The purpose of this study is to develop and test a smoking cessation intervention for persons who are specifically sensitive to anxiety and anxiety-related bodily sensations.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 65 years old
2. Not pregnant
3. Regular smoker averaging 10 or more cigarettes per day for at least one year
4. Score of 25 or greater on 16-item Anxiety Sensitivity Index
5. Motivation to Quit score of 7 or greater (using Readiness to Quit Ladder)
6. Not currently using pharmacotherapy for smoking cessation (e.g., Zyban)
7. No use of other tobacco products (e.g., chewing tobacco, cigars)
8. No Axis-I or Axis-II diagnoses other than mood or anxiety disorders (intake interview required)
9. No suicidal or homicidal ideation
10. No current psychotropic medication use
11. No evidence of substance abuse or dependence (other than nicotine dependence)
12. No history of significant medical conditions (cardiovascular, neurological, etc.)
13. Ability to provide informed, written consent (no evidence of limited mental capacity)
14. Sufficient command of the English language (able to carry on interview conversation)
15. Plan to stay in Burlington VT area for at least next 6 months

Exclusion Criteria:

1. Not between 18-65 years old
2. Pregnant or currently trying to become pregnant
3. Regular smoker for less than one year OR smoke less than 10 cigarettes per day
4. ASI below cutoff level of 25
5. Motivation to Quit score of 6 or less (using Readiness to Quit Ladder)
6. Current or recent use of any pharmacotherapy for smoking cessation (e.g., patch, Zyban)
7. Current use of other tobacco products (e.g., chewing tobacco, cigars)
8. Axis-I disorders other than anxiety or mood disorders.
9. Endorsement of suicidality or homicidal ideation.
10. Any current psychotropic medication use (must have stopped at least 1 month prior).
11. Any evidence of substance abuse or dependence (other than nicotine dependence)
12. Any history of significant medical conditions (cardiovascular, neurological, etc.)
13. Inability to provide informed, written consent (evidence of limited mental capacity)
14. Insufficient command of the English language (unable to carry on conversation)
15. Plan to permanently leave Burlington area anytime during the next 6-12 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2005-01; Primary Completion 2009-08 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Smoking status | 2 weeks post Quit Day
Smoking status | 4 weeks post Quit Day
Smoking status | 8 weeks post Quit Day
Smoking status | 16 weeks post Quit Day
Smoking status | 24 weeks post Quit Day

SECONDARY OUTCOMES:
Where applicable, length of time from Quit Day to relapse. | Determined at conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Zvolensky, Ph.D., Principal Investigator — University of Vermont, Department of Psychology; Andrew R. Yartz, Ph.D., Study Director — University of Vermont, Department of Psychology
Locations (1):
- University of Vermont, Burlington, Vermont, United States